CLINICAL TRIAL: NCT01246323
Title: Combined General and Spinal Anesthesia vs. General Anesthesia for Pain Relief During Laparoscopy Gynecological Surgery
Brief Title: Combined Anesthesia for Laparoscopy Surgery in Gynecology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Lior Lowenstein, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COBINED ANASTHESIA GYNECOLOGY
Record Dates: First submitted 2010-11-14; First posted 2010-11-23 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2010-11

CONDITIONS: Pain
Keywords: Visual analogue scale; pain level; analgesia; combined anesthesia
MeSH Terms: conditions — Pain; Agnosia | interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- combined anesthesia (Active Comparator): Patients will receive spinal and general anesthesia for benign laparoscopy gynecological surgery
  Interventions: Procedure: Spinal anesthesia with Fentanyl+ Morphine
- Control (No Intervention)

INTERVENTIONS:
Procedure: Spinal anesthesia with Fentanyl+ Morphine — Fentanyl 15 microgram Morphine 0.1-0.5 mg
  Arms: combined anesthesia

SUMMARY:
The purpose of this study is to determine whether combined anesthesia will provide better pain control for the postoperative period following gynecological laparoscopy surgery.

DETAILED DESCRIPTION:
Following signing an informed consent patients who are scheduled for gynecological laparoscopy surgery for benign disease will randomized to general vs. combined general and spinal anesthesia.

During the postoperative period data regarding pain level as evaluated by visual analogue scale (VAS), number of doses of pain relief drugs, satisfaction and number of day in hospitalization will be collected from patient charts.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiology (ASA) physical status classification system:ASA I-III.
2. Benign Gynecological Laparoscopy surgery

Exclusion Criteria:

1. Patients who are not capable to sign the consent form.
2. Women with known allergy to the medication used in spinal analgesia.
3. Patients who are pregnant or lactating.
4. Patients with contraindication to spinal analgesia.
5. Patients who use opioid on a regular base.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-11 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Pain level | For the first 72 hours following surgery
  Pain level will be evaluated every 4 hours from the time of surgery to discharge
Number of doses of analgesic drugs | For the first 72 hours following surgery
  Number of doses of analgesic medications will be collected from patients charts.

CONTACTS AND LOCATIONS:
Overall Officials: Lior Lowenstein, Study Chair — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

REFERENCES:
- [Background] Jones T, Tilsley DW, Wilson CB, Lammertsma AA, Brown G, Brady F, Price PM. Positron emission tomography for tumour assessment. NMR Biomed. 1992 Sep-Oct;5(5):265-9. doi: 10.1002/nbm.1940050512. PMID 1449966
- [Background] Motamed C, Bouaziz H, Franco D, Benhamou D. Analgesic effect of low-dose intrathecal morphine and bupivacaine in laparoscopic cholecystectomy. Anaesthesia. 2000 Feb;55(2):118-24. doi: 10.1046/j.1365-2044.2000.055002118.x. PMID 10651671
- [Background] Kong SK, Onsiong SM, Chiu WK, Li MK. Use of intrathecal morphine for postoperative pain relief after elective laparoscopic colorectal surgery. Anaesthesia. 2002 Dec;57(12):1168-73. doi: 10.1046/j.1365-2044.2002.02873.x. PMID 12437707
- [Background] Karaman S, Kocabas S, Uyar M, Zincircioglu C, Firat V. Intrathecal morphine: effects on perioperative hemodynamics, postoperative analgesia, and stress response for total abdominal hysterectomy. Adv Ther. 2006 Mar-Apr;23(2):295-306. doi: 10.1007/BF02850135. PMID 16751162